CLINICAL TRIAL: NCT00161902
Title: A Randomized, Controlled, Multicenter Study to Evaluate Efficacy and Safety of Fibrin Sealant VH S/D for Hemostasis in Subjects Undergoing Total Hip Replacement
Brief Title: Efficacy and Safety of Fibrin Sealant Vapor Heated Solvent/Detergent Treated (FS VH S/D) for Hemostasis in Subjects Undergoing Total Hip Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 550001
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Hip Replacement Surgery
Keywords: Arthroplasty; Hip Prosthesis; Cement Free Hip Prosthesis; Femur Head Necrosis; Coxarthrosis
MeSH Terms: conditions — Femur Head Necrosis; Osteoarthritis, Hip

INTERVENTIONS:
Drug: Fibrin Sealant Vapor-Heated Solvent/Detergent-treated

SUMMARY:
The purpose of the study is to monitor the safety of FS VH S/D and evaluate whether FS VH S/D is superior to standard treatment in reducing blood loss in subjects undergoing total hip replacement with cement-free hip prostheses.

ELIGIBILITY:
Inclusion Criteria:

Each subject to be included into the study must fulfill the following inclusion criteria:

* Subjects receiving a cement free hip prosthesis due to coxarthrosis because of primary or dysplastic arthrosis grade 1 - 3 according to Crowe or rheumatoid arthritis as well as subjects receiving a cement free hip prosthesis due to femur head necrosis (Crowe classification).
* ASA and NSAIDs have been discontinued one week prior to surgery
* Written informed consent
* Male and female at least 19 years of age

Exclusion Criteria:

Subjects fulfilling the following exclusion criteria will not be recruited into the study:

* Impaired coagulation
* Previous hip surgery
* Acetabular roof plastic
* Known hypersensitivity to aprotinin or other components of the product
* Immunodeficiency
* Increased red cell production
* Pregnant or lactating women (positive urine or serum pregnancy test; this test is required of any female subject who is not post menopausal or surgically sterilized).
* Subjects concurrently participating in another clinical trial or having received another investigational drug within the last 30 days.

Also patients with abnormal coagulation values due to anticoagulants like coumadins or heparin must be excluded.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Florian Gottsauner-Wolf, MD, Principal Investigator — A. ö. Krankenhaus Krems, Austria; Axel Rüter, MD, Principal Investigator — Klinik für Unfall- und Wiederherstellungschirurgie des Zentralklinikums Augsburg, Germany
Locations (7):
- Austria (3):
  - A. ö. Krankenhaus Krems, Abteilung f. Orthopädie, Krems, Lower Austria
  - Allgemeines Krankenhaus der Stadt Wien, University Clinic for Orthopedics, Vienna
  - Donauspital im SMZ Ost, Department of Orthopedic Surgery, Vienna
- Klinik für Unfall- u. Wiederherstellungschirurgie des Zentralklinikums Augsburg, Augsburg, Germany
- Netherlands (3):
  - St. Anna Ziekenhuis, Orthopedic Surgery, Geldrop
  - Academisch Ziekenhuis Maastricht, Orthopedic Surgery, Maastricht
  - St. Clara Ziekenhuis, Orthopedic Surgery, Rotterdam